CLINICAL TRIAL: NCT03150225
Title: The Impact of Physical Exercise on Androgen Deficiency of Male Aging in Physical, Psychological, Hormonal and Sexual Aspects: a Randomized Clinical Trial
Brief Title: Physical Exercise for Men With Andropause
Acronym: DAEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratório de Pesquisa em Lazer e Atividade Física (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.011.641
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Androgen Deficiency; Depressive Symptoms; Stress, Psychological; Abdominal Obesity; Testosterone Deficiency; Erectile Dysfunction
Keywords: andropause; depressive symptoms; stress; abdominal Obesity; testosterone; erectile dysfunction
MeSH Terms: conditions — Depression; Stress, Psychological; Obesity, Abdominal; Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: The randomization of the men who will participate in the study will be carried out through a computer program; In the four groups that will compose the study: exercise group + supplementation - intervention with application of a concurrent training protocol for six months and supplementation with eurycoma longifolia, 200mg once daily; exercise group + placebo intervention with application of a concurrent training protocol for six months and administration of starch capsules; control group + supplementation - monthly will be contacted via telephone and will be encouraged to maintain their daily activities and supplementation with eurycoma longifolia, 200mg once daily; control group + placebo - monthly will be contacted via telephone and will be encouraged to maintain their daily activities and administration of starch capsules.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will have a double-blind blindness, performed in the process of randomization of the participants, who will not be informed about the allocation of the groups, and in the period of data collection and application of the concurrtent training protocol, in which the Researchers who will carry out the data collection will not participate in the application of the protocol, and vice versa.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise group + supplementation (Experimental): It will be composed of participants randomly assigned to this group, reinforcing the importance of attendance in classes (minimum of 75% of frequency) for significant health benefits. The evaluation measures will be made through a self-administered questionnaire and physical evaluations (cardiorespiratory fitness, body mass index, percentage of fat, waist circumference and muscular strength). The intervention with the concurrent training will be carried out in a gymnasium in Florianópolis, Santa Catarina. After all the evaluation procedures have been performed, the intervention period will begin, being three times a week, lasting 60 minutes, according to the study protocol.
  In addition participants will receive supplementation of Eurycoma longifolia in 200mg capsules with standardized extract in aqueous-soluble extract and should be taken daily.
  Interventions: Other: Concurrent training; Dietary Supplement: Eurycoma longifolia
- Control group + supplementation (Active Comparator): Will be reinforced to the participants of this group the importance of maintaining their daily activities. In addition participants will receive supplementation of Eurycoma longifolia in 200mg capsules with standardized extract in aqueous-soluble extract and should be taken daily.
  Interventions: Dietary Supplement: Eurycoma longifolia
- Exercise group + placebo (Experimental): It will be composed of participants randomly assigned to this group, reinforcing the importance of attendance in classes (minimum of 75% of frequency) for significant health benefits. The evaluation measures will be made through a self-administered questionnaire and physical evaluations (cardiorespiratory fitness, body mass index, percentage of fat, waist circumference and muscular strength). The intervention with the concurrent training will be carried out in a gymnasium in Florianópolis, Santa Catarina. After all the evaluation procedures have been performed, the intervention period will begin, being three times a week, lasting 60 minutes, according to the study protocol.
  In addition participants will receive starch capsules to be taken daily.
  Interventions: Other: Concurrent training
- Control group + placebo (No Intervention): Will be reinforced to the participants of this group the importance of maintaining their daily activities. In addition participants will receive starch capsules to be taken daily.

INTERVENTIONS:
Other: Concurrent training — In this protocol the participants will perform aerobic and resistance training according to published evidence for middle-aged men; Characterized as concurrent training.
  The protocol will last six months and will be divided into two quarters. In the first trimester, initial 30 minutes will be assigned to resistance training, followed by 30 minutes of aerobic training; Already in the second trimester will be 20 initial minutes for the aerobic training and later 40 minutes for the resistance training; Aiming to obtain benefits in the levels of muscular strength, aerobic capacity, body composition, besides positive results in relation to the hormonal adaptations of testosterone, as well as in the psychological well being of the participants. Classes will occur at a frequency of three times weekly, lasting 60 minutes a session.
  Arms: Exercise group + placebo; Exercise group + supplementation
Dietary Supplement: Eurycoma longifolia — Eurycoma longifolia will be administered by supplementation with the standard aqueous-soluble extract extract (Physta ™) in single 200mg capsules daily, and placebo by starch capsules. The supplementatio will last six months.
  Arms: Control group + supplementation; Exercise group + supplementation

SUMMARY:
The aim of this study is to analyze the impact of physical exercise through a protocol of concurrent training in the psychological, physical, hormonal and sexual aspects in middle aged men with androgen deficiency in the aging male (ADAM). The study design with randomized clinical trial, comprising men in middle age (40 to 59 years) with ADAM, should be divided into two groups: 1) Control group (CG); 2) Experimental group (EG). Information related to sociodemographic and clinical profile will be collected; Psychological aspects (depressive and anxiety symptoms - Hospital Anxiety and Depression Scale ; stress - Perceived Stress Scale); Physical acpects (IMC; Percentage of body fat; Abdominal obesity - waist circumference in cm; Muscle strength - Biodex System 4 PRO isokinetic dynamometer; cardiorespiratory Fitness - Cycle-ergometer - CASE ECG Stress Testing System, General Electric Medical Systems, Milwaukee, WI); Hormonal aspects (total and free testosterone - blood collection); Sexual Aspect (Sexual satisfaction- International Index of Erectile Function); DAEM (scale of symptoms of aging). Apply a physical exercise protocol using the functional training method over a six-month period. All information will be collected before and after the intervention period. For statistical analysis, use the SPSS statistical package, version 20.0. (Kolmogorov-Smirnov or Shapiro-Wilk test) for the selection of statistical tests.

DETAILED DESCRIPTION:
In this protocol the participants will perform aerobic and resistance training according to published evidence for middle-aged men; Characterized as concurrent training.

The protocol will last six months and will be divided into two quarters. In the first trimester, initial 30 minutes will be assigned to resistance training, followed by 30 minutes of aerobic training; Already in the second trimester will be 20 initial minutes for the aerobic training and later 40 minutes for the resistance training; Aiming to obtain benefits in the levels of muscular strength, aerobic capacity, body composition, besides positive results in relation to the hormonal adaptations of testosterone, as well as in the psychological well being of the participants.

Classes will occur at a frequency of three times weekly, lasting 60 minutes a session.

For the elaboration of this protocol will be followed the guidelines of the American College of Sports Medicine of resistance training for healthy adults The aerobic training of this protocol will follow the American College of Sports Medicine's prescription prescription guidelines for the health of healthy adult subjects,

ELIGIBILITY:
Inclusion Criteria:

* men presenting ADAM according to their responses on the Aging Male Symptoms Scale and testosterone levels <220 pmol/l

Exclusion Criteria:

* history of neurological or musculoskeletal diseases or who have prostate cancer will be excluded, as also those who have been submitted toresistance and/or aerobic in the three months prior to data collection

Ages: 40 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Androgen deficiency in the aging male | five minutes
  "AGING MALE SYMPTOMS SCALE" With symptoms, without symptoms; Mild, moderate and severe symptoms

SECONDARY OUTCOMES:
Cardiorespiratory fitness | 10 minutes
  Submaximal ergometric test - Expiratory flow volume
Body mass index | 5 minutes
  Body mass (Kg) divided by the square of the height (m2) - Normal (up to 24.9 Kg/m2), overweight (from 25 Kg/m2 to 29.9 Kg/m2) & obesity (above 30 Kg/m2)
Percent fat | 10 minutes
  Ultrasound (triceps, abdominal and subscapular adipose tissue) - Results in percentage (%)
Waist circumference | 5 minutes
  The waist circumference will be measured at the natural waist level, the mean point between the upper anterior iliac crest and the last rib - Level 1 - increased cardiovascular risk; level 2 - substantially increased cardiovascular risk
Muscle strength | 10 minutes
  Computer based multifunctional dynamometer system - Maximal repetitions
Symptoms of depression | 5 minutes
  BDI - Beck's Depression Inventory - No symptoms of depression, mild symptoms of depression, moderate symptoms of depression, severe symptoms of depression
Stress level | 5 minutes
  Perceived stress scale - The scores can vary from 0 to 56, the nearer to 56 the greater the stress level
Testosterone levels | 5 minutes
  Blood test - Limits below <220 pmol/l (indication of ADAM)
Sexual satisfaction | 10 minutes
  IEFI International Erectile Function Index - Good sexual quality of life Bad sexual quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Melissa CS Vieira, MSc, Principal Investigator — Santa Catarina State University - Florianópolis, SC, Brazil; Adriana CA Guimarães, PhD, Study Director — Santa Catarina State University - Florianópolis, SC, Brazil
Locations (1):
- Santa Catarina State University, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No